

Statistical Analysis: Data analysis was performed using the SPSS 24.0 (IBM Statistics, PASW Inc, Chicago, IL, USA) program. The distribution of data was examined with the Kolmogorov-Smirnov test. Descriptive statistics were presented as numbers, percentages, means, medians, standard deviations, minimum and maximum values. Variables were analyzed using chi-square, ANOVA, and Kruskal-Wallis tests based on their distribution. The Kruskal-Wallis hypothesis test assessed differences between groups in repeated measurements. Scale scores and relationships between positions were evaluated using Simple Linear Regression analysis. The statistical significance threshold was set at p<0.05.

Table 1: Comparison of CGT Positions in terms of Sociodemographic and Obstetric Features

| Variables | | Right<br>Lateral<br>Side-<br>Lying<br>Position | | Semi-<br>Fowler<br>Position | | Left Lateral Side-Lying Position | | Test<br>Score | p |
|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | <u>%</u> | | |
| Age | Below age 18 | 0 | 0.0 | 0 | 0.0 | 2 | 1.6 | | 0.001 |
| $(\overline{X}\pm SD,$ | 19-34 | 42 | 68.9 | 48 | 77.4 | 93 | 78.2 | 3.795** | 0.391*** |
| 31.62±4.46) | 35 and over | 19 | 31.1 | 14 | 22.6 | 24 | 20.2 | | |
| | 18 and below | - | - | - | - | - | - | | |
| | (underweight) | 1.6 | 26.2 | 20 | 22.2 | 31 | 26.1 | | |
| DMI | 19-24 (normal)<br>25-29 | 16 | 20.2 | 20 | 32.3 | 31 | 20.1 | | |
| BMI | | 32 | 52.5 | 28 | 45.2 | 61 | 51.3 | | |
| | (overweight) 30 and over | | | | | | | | |
| | | 13 | 21.3 | 14 | 22.6 | 27 | 22.7 | | |
| | (obese) Officially | | | | | | | | |
| | Married, Partner | 59 | 96.7 | 62 | 100 | 115 | 96.6 | | |
| | in a Civil union | 39 | 90.7 | 02 | 100 | 113 | 90.0 | | 0.375* |
| Civil Status | Partner in a | | | | | | | 2.025** | |
| Civii Status | Civil Union,<br>Not Officially<br>Married | 2 | 3.3 | 0 | 0.0 | 4 | 3.4 | 2.023 | 0.575 |
| | Primary School | 12 | 20.0 | 7 | 11.3 | 22 | 18.6 | | |
| | Middle School | 9 | 15.0 | 15 | 24.2 | 22 | 18.6 | <del>-</del> | |
| | High school | 18 | 30.0 | 19 | 30.6 | 36 | 30.5 | - | |
| | Associate | | | 7 | | 1.1 | | - | |
| Education | Degree | 6 | 10.0 | 7 | 11.3 | 11 | 9.3 | 0.310** | 0.298* |
| | Bachelor's | 11 | 18.3 | 13 | 21.0 | 26 | 22.0 | _' | |
| | Degree | 11 | 18.3 | 13 | 21.0 | 20 | 22.0 | _ | |
| | Graduate | 4 | 6.7 | 1 | 1.6 | 1 | 0.8 | | |
| | Degree | 4 | 0.7 | 1 | 1.0 | 1 | 0.8 | | |
| Employment | Employed | 15 | 25.0 | 12 | 19.4 | 30 | 25.6 | 0.940** | 0.628* |
| Employment | Unemployed | 45 | 75.0 | 50 | 80.6 | 87 | 74.4 | 0.740 | 0.026 |
| Place of | Province | 42 | 73.7 | 56 | 91.8 | 87 | 73.7 | - | |
| Residence | District | 15 | 26.3 | 5 | 8.2 | 29 | 24.6 | 7.285** | 0.004* |
| RUSIMUNICU | Village | 0 | 0.0 | 0 | 0.0 | 2 | 1.7 | | |
| | Income greater | 5 | 8.3 | 3 | 4.8 | 11 | 9.2 | | |
| | than expenditure | | 0.5 | | 1.0 | | | <u>-</u> | |
| Income Level | Income equal to | 34 | 56.7 | 35 | 56.5 | 65 | 54.6 | 0.465** | 0.269* |
| Income Level | expenditure | J. | 30.7 | | | | | - 0.105 | 0.209 |
| | Income less than | 21 | 35.0 | 24 | 38.7 | 43 | 36.1 | | |
| | expenditure | | | | | | | | |
| Social<br>Security? | Yes | 51 | 85.0 | 52 | 85.2 | 99 | 85.3 | 0 00 444 | 0.0004 |
| | No | 9 | 15.0 | 9 | 14.8 | 17 | 14.7 | 0.004** | 0.998* |
| <u> </u> | | | | | | 8 | 6.8 | | |
| Any medical | Yes | 4 | 6.7 | 5 | 8.1 | · · | 0.8 | 0.085** | 0.438* |
| problem? | No | 56 | 93.3 | 57 | 91.9 | 110 | 93.2 | | |
| Prognancy | Planned | 91 | 76.5 | 51 | 82.3 | 91 | 76.5 | 5.825** | 0.054* |
| Pregnancy | Unplanned | 28 | 23.5 | 11 | 17.7 | 28 | 23.5 | 3.023 | 0.034 |

| Wanted | Yes | 54 | 93.4 | 59 | 95.2 | 114 | 958 | 0.086** | 0.446* |
|---|---|---|---|---|---|---|---|---|---|
| Pregnancy? | No | 4 | 6.6 | 3 | 4.8 | 5 | 42 | 0.080 | 0.440 |
| Number of | Primipara | 12 | 20.3 | 21 | 37.5 | 39 | 33.3 | 1 52(** | 0.104 |
| pregnancies | Multipara | 47 | 79.7 | 35 | 62.5 | 78 | 67.7 | 4.536** | 0.104 |
| Ending Week | 36th week or earlier | 31 | 51.7 | 39 | 62.9 | 66 | 55.9 | | |
| of Last | 37th-40th week | 29 | 48.3 | 23 | 37.1 | 49 | 41.5 | 1.085** | 0.167* |
| Pregnancy | 41st week or later | 0 | 0.0 | 0 | 0.0 | 3 | 2.5 | • | |
| Number of | None | 17 | 28.8 | 22 | 39.3 | 46 | 39.3 | | |
| living children | 1-3 | 41 | 69.5 | 34 | 60.7 | 67 | 57.3 | 0.025** | 0.467* |
| iiving children | 4 or more | 1 | 1.7 | 0 | 0.0 | 4 | 3.4 | | |
| Number of | None | 43 | 72.9 | 40 | 72.7 | 101 | 86.3 | | |
| Miscarriages | 1-2 | 15 | 25.4 | 10 | 18.2 | 16 | 13.7 | 9.306** | 0.002* |
| Miscarriages | 3 or more | 1 | 1.7 | 5 | 9.1 | 0 | 0 | | |
| Number of | None | 50 | 86.2 | 46 | 82.1 | 107 | 91.5 | | |
| Wanted | 1-3 | 7 | 12.1 | 10 | 17.9 | 10 | 8.5 | 3.142** | 0.051* |
| Miscarriages | 4 or more | 1 | 1.7 | 0 | 0.0 | 0 | 0.0 | | |
| Mode of | Vaginal delivery | 25 | 45.5 | 16 | 32.7 | 30 | 28.8 | | |
| Delivery in | Cesarean | 21 | 38.2 | 19 | 38.8 | 47 | 45.2 | 5.440** | 0.247* |
| Last<br>Pregnancy | No delivery | 9 | 16.4 | 14 | 28.6 | 27 | 26.0 | 3.440 | 0.247 |
| Position<br>during<br>previous CTG | Left Lateral<br>Side-Lying<br>Position | 41 | 74.5 | 37 | 67.3 | 78 | 79.6 | | |
| | Right Lateral<br>Side-Lying<br>Position | 12 | 21.8 | 9 | 16.4 | 19 | 19.4 | 13.668** | 0.006* |
| * ************************************* | Semi-Fowler<br>Position | 2 | 3.6 | 9 | 16.4 | 1 | 1.0 | | |

\*p<0.05, \*\*Chi-squared analysis

Table 2. Comparison of CTG Evaluation Parameters according to CTG Position

| Variables | CTG<br>Duratio<br>n | Right Lateral<br>Side-Lying<br>Position<br>(1) | | Semi-Fowler<br>Position<br>(2) | | Left Lateral<br>Side-Lying<br>Position<br>(3) | | Test Score | p | Benfer<br>roni<br>Group |
|---|---|---|---|---|---|---|---|---|---|---|
| | | X | SD | Ā | SD | X | SD | | | |
| Starting time of CTG | | 11.76 | 2.14 | 11.30 | 1.87 | 11.76 | 2.13 | 0.991** | 0.373* | |
| Ending time of CTG | | 13.86 | 13.83 | 11.61 | 1.84 | 12.09 | 2.14 | 1.635** | 0.197* | |
| CTG Duration | | 20.24 | 1.99 | 18.46 | 2.82 | 20.25 | 3.07 | 8.919** | 0.000* | 2>1,<br>2>3 |
| | In first 5 minutes | 138.13 | 9.43 | 143.57 | 7.93 | 137.50 | 10.64 | 7.542** | 0.001* | 2>1,<br>2>3 |
| | 6th-10th<br>minutes | 139.54 | 9.63 | 143.69 | 8.09 | 138.16 | 11.48 | 5.321** | 0.006 | 2>3 |
| Basal Heart<br>Rate | 11th-<br>15th<br>minutes | 140.18 | 9.82 | 143.87 | 8.88 | 139.36 | 10.70 | 3.769** | 0.025* | 2>3 |
| | 16th-<br>20th<br>minutes | 140.04 | 9.40 | 143.35 | 8.40 | 139.53 | 10.47 | 2.939** | 0.055* | |
| | In first 5 minutes | 168.33 | 10.40 | 168.75 | 7.50 | 175. | 5.00 | 0.700** | 0.528* | |
| | 6th-10th minutes | 170.00 | 0.00 | 172.00 | 5.70 | 170.00 | 0.00 | 0.205** | 0.820* | |
| Fetal<br>tachycardia | 11th-<br>15th<br>minutes | 168.00 | 0.00 | 170.00 | 5.4 | 172.00 | 4.87 | 1.409** | 0.543* | |
| | 16th-<br>20th<br>minutes | 165.00 | 0.00 | 170.00 | 5.00 | 175.00 | 7.07 | 1.063** | 0.448* | |
| | At 5th minute | - | - | - | - | - | - | - | - | |
| Bradycardia | 6th-10th<br>minutes | 100.00 | - | 107.50 | 10.60 | - | - | 0.333 | 0.667* | |
| | 11th-<br>15th<br>minutes | - | - | - | - | - | - | - | - | |
| | 16th-<br>20th<br>minutes | - | - | - | - | - | - | - | - | |
| | In first 5 minutes | 4.80 | 4.07 | 3.72 | 2.34 | 7.48 | 5.22 | 15.980** | 0.000* | 3>2,<br>3>1 |
| | 6th-10th<br>minutes | 4.54 | 3.98 | 3.55 | 2.71 | 6.58 | 5.55 | 9.100** | 0.000* | 3>2,<br>3>1 |
| Fetal<br>Movement | 11th-<br>15th<br>minutes | 4.49 | 3.72 | 3.05 | 2.46 | 6.49 | 4.87 | 13.829** | 0.000* | 3>2,<br>3>1 |
| | 16th-<br>20th<br>minutes | 4.39 | 3.95 | 3.05 | 2.21 | 6.52 | 4.33 | 16.720** | 0.000* | 3>2,<br>3>1 |
| Number of | In first 5 minutes | 2.96 | 3.14 | 2.74 | 2.53 | 2.95 | 2.88 | 0.442*** | 0.802 | |
| Contractions | 6th-10th<br>minutes | 1.93 | 2.70 | 1.90 | 2.63 | 1.69 | 2.28 | 0.151*** | 0.927* | |

| | 11th-<br>15th<br>minutes | 1.09 | 0.396 | 0.98 | 0.23 | 1.12 | 0.376 | 5.835*** | 0.054* | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 16th-<br>20th<br>minutes | 1.16 | 0.77 | 1.32 | 1.05 | 1.08 | .056 | 1.313*** | 0.519* | |
| Intensity of<br>Contraction | In first 5 minutes | 26.31 | 24.34 | 20.23 | 22.86 | 25.06 | 24.23 | 1.011*** | 0.603 | |
| | 6th-10th<br>minutes | 46.16 | 23.54 | 44.98 | 22.18 | 46.28 | 21.60 | 0.028*** | 0.986* | |
| | 11th-<br>15th<br>minutes | 46.16 | 23.54 | 44.98 | 22.18 | 46.28 | 23.54 | 0.028*** | 0.986* | |
| | 16th-<br>20th<br>minutes | 25.75 | 10.34 | 22.26 | 20.00 | 24.82 | 10.54 | 0.102 | 0.950* | |
| | In first 5 minutes | 1.08 | 1.03 | 1.61 | 1.05 | 1.11 | 0.96 | 5.318** | 0.006* | 2>1,<br>2>3 |
| | 6th-10th minutes | 1.18 | 1.08 | 1.51 | 1.11 | 1.18 | 1.08 | 2.015** | 0.136* | |
| Accelerations | 11th-<br>15th<br>minutes | 1.39 | 1.14 | 1.74 | 1.10 | 1.40 | 1.08 | 1.953** | 0.144* | |
| | 16th-<br>20th<br>minutes | 1.32 | 1.22 | 1.70 | 1.50 | 1.45 | 1.12 | 1.347** | 0.262* | |
| | In first 5 minutes | 0.06 | 0.24 | 0.11 | 0.46 | 0.18 | 0.55 | 1.895*** | 0.388* | |
| Decelerations | 6th-10th<br>minutes | 0.04 | 0.21 | 0.21 | 0.68 | 0.27 | 0.62 | 8.075** | 0.018* | 1>3 |
| | 11th-<br>15th<br>minutes | 0.08 | 0.33 | 0.12 | 0.38 | 0.15 | 0.40 | 2.255*** | 0.324* | |
| | 16th-<br>20th<br>minutes | 0.04 | 0.21 | 0.07 | 0.26 | 0.18 | 0.50 | 4.439*** | 0.109* | |

<sup>\*</sup>p<0.005, \*\* Anova test, \*\*\*Kruskal Wallis Test

**Table 3: Intergroup Comparison of Vital Signs During CTG** 

| | | Right Lateral Side-Lying Position (1) $\bar{X} \pm SD$ | Semi-<br>Fowler<br>Position<br>(2)<br>$\bar{X} \pm SD$ | Left Lateral Side- Lying Position (3) $\bar{X} \pm SD$ | Test Score | р | Benfe<br>rroni<br>Grou<br>p | Benferr<br>oni<br>Time |
|---|---|---|---|---|---|---|---|---|
| Blood<br>Pressure<br>(Systolic) | Before CTG (1) At the mome nt of CTG (2) After CTG (3) | 113.67±10.<br>06<br>110.37±9.4<br>1<br>115.91±10.<br>76 | 108.16±10.<br>56<br>107.00±8.5<br>7<br>100.08±8.1<br>5 | 112.80±1<br>1.21<br>108.89±1<br>1.00<br>113.56±1<br>2.28 | $F_{Group} = 7.964$ $F_{Time} = 13.014$ $F_{GroupxTime} = 2.649$ | 0.000*<br>0.000*<br>0.000* | 2>3,<br>2>1 | 1>3, 1>2 |
| Blood<br>Pressure<br>(Diastolic) | Before CTG (1) At the mome nt of CTG (2) After CTG (3) | 71.00±9.06<br>67.00±9.60<br>70.41±10.1<br>8 | 66.83±6.83<br>64.29±7.26<br>64.64±7.29 | 69.20±9.9<br>0<br>66.56±11.<br>70<br>71.10±11.<br>36 | $F_{Group} = 6.829$ $F_{Time} = 9.940$ $F_{GroupxTime} = 2.049$ | <b>0.000* 0.000*</b> 0.090* | 1>3,<br>1>2 | 2=3>1 |
| Pulse | Before CTG (1) At the mome nt of CTG (2) After CTG (3) | 94.70±10.8<br>4<br>92.24±10.6<br>0<br>92.06±10.5<br>3 | 97.77±11.0<br>3<br>95.88±10.5<br>1 | 93.37±12.<br>28<br>89.84±11.<br>29<br>91.77±10.<br>23 | $F_{Group} = 5.461$ $F_{Time} = 10.315$ $F_{GroupxTime} = 0.822$ | <b>0.005</b> * <b>0.000</b> * 0.512* | 2>1,<br>2>3 | 3>2,<br>2>1 |
| Body<br>Temperat<br>ure | Before CTG (1) At the mome nt of CTG (2) After CTG (3) | 36.32±0.46<br>36.40±0.50<br>36.41±0.49 | 36.29±0.15<br>36.26±0.17<br>36.24±0.14 | 36.49±0.4<br>9<br>36.60±0.5<br>1<br>36.58±0.5 | $F_{Group}=11.77$ $6$ $F_{Time}=3.975$ $F_{GroupxTime}=$ $3.232$ | 0.000*<br>0.023*<br>0.015* | 3>2,<br>3>1 | 1>2>3 |

Table 4. Comparison of Effect of Body Mass Index on CTG Position and Vital Signs

| | Group | $\overline{X}$ | SD | F | р | Bonferroni |
|---|---|---|---|---|---|---|
| G 4 P | Right Lateral<br>Side-Lying<br>Position (1) | 115.91 | 10.76 | | | |
| Systolic<br>Blood | Semi-Fowler<br>Position (2) | 107.08 | 8.15 | 26.785** | 0.002* | 2>3, 1>3 |
| Pressure - | Left Lateral Side-Lying Position (3) | 113.56 | 12.28 | _ | | |
| BMI | | | | 2.734** | 0.157 | |
| Group*BMI <sup>1</sup> | | | | 0.323** | 0.862 | |
| Diastolic | Right Lateral<br>Side-Lying<br>Position (1) | 70.41 | 10.18 | _ | | |
| Blood<br>Pressure | Semi-Fowler<br>Position (2) | 64.64 | 7.29 | 14.054** | 0.010* | 2>3, 2>1 |
| Tressure | Left Lateral<br>Side-Lying<br>Position (3) | 71.10 | 11.36 | | | |
| BMI | | | | 2.193** | 0.214 | |
| Group*BMI | | | | 0.518** | 0.722 | |
| | Right Lateral<br>Side-Lying<br>Position (1) | 92.06 | 10.53 | _ | | |
| Pulse | Semi-Fowler Position (2) | 96.20 | 9.31 | 6.002** | 0.053 | - |
| | Left Lateral<br>Side-Lying<br>Position (3) | 91.77 | 10.23 | | | |
| BMI | | | | 0.461** | 0.658 | |
| Group*BMI | | | | 0.733** | 0.570 | |
| | Right Lateral<br>Side-Lying<br>Position (1) | 36.41 | 0.49 | _ | | |
| Body<br>Temperature | Semi-Fowler<br>Position (2) | 36.24 | 0.14 | 88.070** | 0.000* | 2>3 |
| | Left Lateral<br>Side-Lying<br>Position (3) | 36.58 | 0.51 | | | |
| BMI | | | | 3.572** | 0.072 | |
| Group*BMI | BMI: Body Mass Index | | | 0.076** | 0.989 | |

\*p<0.05 \*\* Ancova, <sup>1</sup>BMI: Body Mass Index

Table 5. Effect of CTG Position on General Comfort Questionnaire Score

| Dependent<br>Variable | Independent<br>Variable | β | Standard<br>Error | Beta | t | p | F | Model (p) | R2 |
|---|---|---|---|---|---|---|---|---|---|
| | (Constant) | 3.398 | 0.168 | - | 20.168 | 0.000* | | | |
| | Right Lateral<br>Side-Lying<br>Position | 163 | 0.094 | 112 | -1.742 | 0.083 | 3.034 | 0.083 | 0.012 |
| General | (Constant) | 2.506 | 0.163 | - | 15.335 | 0.000* | | | |
| Comfort<br>Questionnaire | Semi-Fowler<br>Position | 0.349 | 0.911 | 0.240 | 3.834 | 0.000* | 14.700 | 0.000* | 0.058 |
| Score | (Constant) | 3.329 | 0.129 | - | 25.786 | 0.000* | | | |
| | Left Lateral<br>Side-Lying<br>Position | 0.143 | 0.081 | 0.113 | -1.758 | 0.080 | 3.090 | 0.080 | 0.013 |

<sup>\*</sup>p<0.05 \*\* Simple Linear Regression